CLINICAL TRIAL: NCT00451451
Title: A Randomized, Multicenter, Placebo-Controlled and Active Reference (Glatiramer Acetate) Comparison Study to Evaluate the Efficacy and Safety of BG00012 in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Efficacy and Safety Study of Oral BG00012 With Active Reference in Relapsing-Remitting Multiple Sclerosis
Acronym: CONFIRM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109MS302
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: relapsing; multiple sclerosis; oral; remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Recurrence; Multiple Sclerosis | interventions — Dimethyl Fumarate; Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BG00012 240 mg Twice Daily (BID) (Experimental): Participants received two 120 mg BG00012 capsules orally twice daily (BID) and two placebo capsules orally once daily (QD)
  Interventions: Drug: BG00012; Drug: Placebo
- BG00012 240 mg 3 Times Daily (TID) (Experimental): Participants received two 120 mg BG00012 capsules orally three times daily (TID)
  Interventions: Drug: BG00012
- Placebo (Placebo Comparator): Participants received two placebo capsules orally three times daily (TID)
  Interventions: Drug: Placebo
- Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD) (Active Comparator): Participants received glatiramer acetate (GA) 20 mg subcutaneous injection once daily (QD)
  Interventions: Drug: Glatiramer Acetate

INTERVENTIONS:
Drug: BG00012
  Other Names: dimethyl fumarate; Tecfidera®
  Arms: BG00012 240 mg 3 Times Daily (TID); BG00012 240 mg Twice Daily (BID)
Drug: Placebo
  Arms: BG00012 240 mg Twice Daily (BID); Placebo
Drug: Glatiramer Acetate
  Arms: Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD)

SUMMARY:
To determine if treatment with BG00012 can decrease the number of MS relapses during a certain time period. Other goals of the study are to determine if, over time, BG00012 treatment can decrease the number of certain types of brain lesions commonly seen in MS patients and slow down the time it takes for MS to get worse.

Other objectives of the study are to determine the safety and tolerability of BG00012, as well as the effect it may have on tests and evaluations used to assess MS. Additionally, glatiramer acetate is being used to compare its benefits and risks with placebo and BG00012.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic disease of the central nervous system that affects approximately 400,000 persons in North America and 365,000 persons in Europe. It is predominantly a disease of young adults, primarily women, with disease onset typically occurring between the ages of 20 and 40.

ELIGIBILITY:
Unless otherwise specified, to be eligible to participate in this study, candidates must meet the following eligibility criteria at the time of the randomization:

Key Inclusion Criteria:

* Must have confirmed diagnosis of RRMS according to McDonald criteria #1-4
* Must have a baseline EDSS between 0.0 and 5.0, inclusive.
* Must have relapsing-remitting disease course.

Key Exclusion Criteria:

* Other chronic disease of immune system, malignancies, urologic, pulmonary, gastrointestinal disease
* Pregnant or nursing women

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1417 (Actual)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (194):
- United States (72):
  - Research Site, Birmingham, Alabama
  - Research Site, Cullman, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Research Site, Loma Linda, California
  - Research Site, Pasadena, California
  - Research Site, Sacramento, California
  - Research Site, Walnut Creek, California
  - Research Site, Boulder, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Meridan, Idaho
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Clinton Township, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Dover, New Hampshire
  - Research Site, Lebanon, New Hampshire
  - Research Site, Freehold, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Amherst, New York
  - Research Site, Buffalo, New York
  - Research Site, Cedarhurst, New York
  - Research Site, Mineola, New York
  - Research Site, Patchogue, New York
  - Research Site, Plainview, New York
  - Research Site, Staten Island, New York
  - Research Site, Stony Brook, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bellevue, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Souderton, Pennsylvania
  - Research Site, Cordova, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Belarus (3):
  - Research Site, Homyel
  - Research Site, Minsk
  - Research Site, Vitebsk
- Belgium (3):
  - Research Site, Lommel
  - Research Site, Sijsele-Damme
  - Research Site, Woluwe
- Bosnia and Herzegovina (3):
  - Research Site, Tuzla, B&H Federation
  - Research Site, Banja Luka, Republic Srpska
  - Research Site, Sarajevo B&H Federation
- Bulgaria (5):
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
- Canada (4):
  - Research Site, Edmonton
  - Research Site, London
  - Research Site, Montreal
  - Research Site, Osijek
- Research Site, San José, Costa Rica
- Croatia (2):
  - Research Site, Rijeka
  - Research Site, Zagreb
- Czechia (3):
  - Research Site, Ostrava
  - Research Site, Ostrava-Moravska
  - Research Site, Prague
- Estonia (4):
  - Research Site, Kuressaare
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
- France (7):
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nîmes
  - Research Site, Strasbourg
- Germany (17):
  - Research Site, Bamberg
  - Research Site, Bayreuth
  - Research Site, Berg Starnberger
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Düsseldorf
  - Research Site, Erbach im Odenwald
  - Research Site, Erlangen
  - Research Site, Giessen
  - Research Site, Halle
  - Research Site, Hanburg
  - Research Site, Heidelberg
  - Research Site, Magdeburg
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Schwerin
- Greece (4):
  - Research Site, Athens
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- India (14):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Calicut
  - Research Site, Chandigarh
  - Research Site, Chennai
  - Research Site, Coimbatore
  - Research Site, Kochi
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Ludhiana
  - Research Site, Mangalore
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Pune
- Ireland (3):
  - Research Site, Cork
  - Research Site, Dublin
  - Research Site, Galway
- Israel (2):
  - Research Site, Holon
  - Research Site, Safed
- Research Site, Riga, Latvia
- Mexico (8):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Morelia, Michoacán
  - Research Site, Monterrey, Nuevo León
  - Research Site, Aguascalientes
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterray
- Research Site, Chisinau, Moldova
- Research Site, Hamilton, New Zealand
- Research Site, Skopje, North Macedonia
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Guaynabo, Puerto Rico
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Târgu Mureş
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
- Slovakia (2):
  - Research Site, Košice
  - Research Site, Martin
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Córdoba
  - Research Site, Gandia
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago de Compostela
  - Research Site, Seville
- Ukraine (7):
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Simferopol
  - Research Site, Zaporizhzhya

REFERENCES:
- [Derived] Amezcua L, Mao-Draayer Y, Vargas WS, Farber R, Schaefer S, Branco F, England SM, Belviso N, Lewin JB, Mendoza JP, Shankar SL; ENDORSE Study Investigators. Efficacy of Dimethyl Fumarate in Young Adults with Relapsing-Remitting Multiple Sclerosis: Analysis of the DEFINE, CONFIRM, and ENDORSE Studies. Neurol Ther. 2023 Jun;12(3):883-897. doi: 10.1007/s40120-023-00475-8. Epub 2023 Apr 15. PMID 37061656
- [Derived] Gold R, Arnold DL, Bar-Or A, Fox RJ, Kappos L, Chen C, Parks B, Miller C. Safety and efficacy of delayed-release dimethyl fumarate in patients with relapsing-remitting multiple sclerosis: 9 years' follow-up of DEFINE, CONFIRM, and ENDORSE. Ther Adv Neurol Disord. 2020 May 12;13:1756286420915005. doi: 10.1177/1756286420915005. eCollection 2020. PMID 32426039
- [Derived] Mehta D, Miller C, Arnold DL, Bame E, Bar-Or A, Gold R, Hanna J, Kappos L, Liu S, Matta A, Phillips JT, Robertson D, von Hehn CA, Campbell J, Spach K, Yang L, Fox RJ. Effect of dimethyl fumarate on lymphocytes in RRMS: Implications for clinical practice. Neurology. 2019 Apr 9;92(15):e1724-e1738. doi: 10.1212/WNL.0000000000007262. Epub 2019 Mar 27. PMID 30918100
- [Derived] Fox RJ, Gold R, Phillips JT, Okwuokenye M, Zhang A, Marantz JL. Efficacy and Tolerability of Delayed-release Dimethyl Fumarate in Black, Hispanic, and Asian Patients with Relapsing-Remitting Multiple Sclerosis: Post Hoc Integrated Analysis of DEFINE and CONFIRM. Neurol Ther. 2017 Dec;6(2):175-187. doi: 10.1007/s40120-017-0077-5. Epub 2017 Aug 2. PMID 28770420
- [Derived] Fernandez O, Giovannoni G, Fox RJ, Gold R, Phillips JT, Potts J, Okwuokenye M, Marantz JL. Efficacy and Safety of Delayed-release Dimethyl Fumarate for Relapsing-remitting Multiple Sclerosis in Prior Interferon Users: An Integrated Analysis of DEFINE and CONFIRM. Clin Ther. 2017 Aug;39(8):1671-1679. doi: 10.1016/j.clinthera.2017.06.012. Epub 2017 Jul 25. PMID 28751099
- [Derived] Fox RJ, Chan A, Zhang A, Xiao J, Levison D, Lewin JB, Edwards MR, Marantz JL. Comparative effectiveness using a matching-adjusted indirect comparison between delayed-release dimethyl fumarate and fingolimod for the treatment of multiple sclerosis. Curr Med Res Opin. 2017 Feb;33(2):175-183. doi: 10.1080/03007995.2016.1248380. Epub 2016 Nov 10. PMID 27733070
- [Derived] Gold R, Giovannoni G, Phillips JT, Fox RJ, Zhang A, Marantz JL. Sustained Effect of Delayed-Release Dimethyl Fumarate in Newly Diagnosed Patients with Relapsing-Remitting Multiple Sclerosis: 6-Year Interim Results From an Extension of the DEFINE and CONFIRM Studies. Neurol Ther. 2016 Jun;5(1):45-57. doi: 10.1007/s40120-016-0042-8. Epub 2016 Mar 1. PMID 26932146
- [Derived] Giovannoni G, Gold R, Fox RJ, Kappos L, Kita M, Yang M, Sarda SP, Zhang R, Viglietta V, Havrdova E. Relapses Requiring Intravenous Steroid Use and Multiple-Sclerosis-related Hospitalizations: Integrated Analysis of the Delayed-release Dimethyl Fumarate Phase III Studies. Clin Ther. 2015 Nov 1;37(11):2543-51. doi: 10.1016/j.clinthera.2015.09.011. Epub 2015 Oct 31. PMID 26526385
- [Derived] Fox RJ, Kita M, Cohan SL, Henson LJ, Zambrano J, Scannevin RH, O'Gorman J, Novas M, Dawson KT, Phillips JT. BG-12 (dimethyl fumarate): a review of mechanism of action, efficacy, and safety. Curr Med Res Opin. 2014 Feb;30(2):251-62. doi: 10.1185/03007995.2013.849236. Epub 2013 Oct 22. PMID 24131282
- [Derived] Fox RJ, Miller DH, Phillips JT, Hutchinson M, Havrdova E, Kita M, Yang M, Raghupathi K, Novas M, Sweetser MT, Viglietta V, Dawson KT; CONFIRM Study Investigators. Placebo-controlled phase 3 study of oral BG-12 or glatiramer in multiple sclerosis. N Engl J Med. 2012 Sep 20;367(12):1087-97. doi: 10.1056/NEJMoa1206328. PMID 22992072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized at 205 investigational sites in 28 countries.
Pre-assignment Details: From screening, 1430 eligible subjects were equally randomized. Of these, 1417 subjects received at least one dose of study treatment and comprised the intent-to-treat (ITT) and safety populations.
Period: Overall Study
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD)
Started | 363 (363 participants were dosed; 363 participants were randomized) | 359 (359 participants were dosed; 362 participants were randomized) | 345 (345 participants were dosed; 345 participants were randomized) | 350 (350 participants were dosed; 360 participants were randomized)
Completed | 278 | 284 | 273 | 292
Not Completed | 85 | 75 | 72 | 58
Not completed — Adverse Event | 11 | 21 | 26 | 10
Not completed — Lost to Follow-up | 11 | 9 | 8 | 11
Not completed — Consent Withdrawn | 14 | 9 | 17 | 17
Not completed — Investigator Decision | 6 | 2 | 1 | 2
Not completed — Subject Non-Compliance | 8 | 4 | 3 | 3
Not completed — Death | 1 | 0 | 0 | 1
Not completed — Other Reasons for Not Completing Study | 34 | 30 | 17 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD) | Total
Number analyzed (Participants) | 363 | 359 | 345 | 350 | 1417
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (9.24) | 37.8 (9.35) | 37.8 (9.39) | 36.7 (9.06) | 37.3 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 245 | 250 | 247 | 993
  Male | 112 | 114 | 95 | 103 | 424
Mean Expanded Disability Status Scale (EDSS) score [Mean (Standard Deviation); unit: units on a scale] — The EDSS scores range from 0.0 (normal exam) to 10.0 (death due to MS).
  units on a scale | 2.59 (1.170) | 2.56 (1.202) | 2.52 (1.185) | 2.57 (1.223) | 2.56 (1.194)
Mean number of relapses within the previous 3 years [Mean (Standard Deviation); unit: Number of relapses] | 2.5 (1.46) | 2.4 (1.27) | 2.6 (1.50) | 2.4 (1.32) | 2.5 (1.39)
Mean number of relapses within the past 12 months [Mean (Standard Deviation); unit: Number of relapses] | 1.4 (0.80) | 1.3 (0.63) | 1.4 (0.72) | 1.4 (0.64) | 1.4 (0.70)
Time since first multiple sclerosis (MS) diagnosis [Mean (Standard Deviation); unit: years] | 4.8 (5.01) | 4.9 (5.11) | 4.6 (5.23) | 4.4 (4.70) | 4.7 (5.01)
Mean number of Gadolinium(Gd)-enhancing T1-weighted lesions [Mean (Standard Deviation); unit: Number of Gd enhancing lesions] — This baseline measure could only be assessed in the magnetic resonance imaging (MRI) cohort. The MRI cohort included 681 intent-to-treat (ITT) subjects who were enrolled at sites that participated in the MRI portion of the study and who had MRI data (167 placebo, 169 BG00012 BID, 170 BG00012 TID, and 175 GA). Sites could participate only if their MRI capability was validated by the independent MRI reading center. Approximately 95% of all subjects enrolled at MRI sites participated in the MRI portion of the study.
  Number of Gd enhancing lesions | 2.7 (7.71) | 2.7 (6.22) | 1.9 (5.02) | 2.4 (6.81) | 2.4 (6.51)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate
Description: A protocol-defined relapse was defined as new or recurrent neurologic symptoms not associated with fever or infection that lasted at least 24 hours, and were separated by at least 30 days from onset of a preceding relapse. All protocol-defined relapses were evaluated by an independent neurologic evaluation committee.
  The adjusted annualized relapse rate was calculated from a negative binomial regression model , adjusted for baseline Expanded Disability Status Scale (EDSS ) score(≤2.0 versus>2.0), age (<40 versus ≥40 years), region, and the number of relapses in the 1 year prior to enrollment.
Time Frame: 2 years
Population: The intent-to-treat (ITT) population was defined as all subjects who were randomized and received at least 1 dose of study treatment. Among subjects who switched to an alternative therapy for multiple sclerosis, all the data before the switch were used for the analysis. In all other subjects, all relapses were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Relapses Per Year
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD)
Number analyzed (Participants) | 363 | 359 | 345 | 350
Relapses Per Year | 0.401 [0.329 to 0.488] | 0.224 [0.179 to 0.282] | 0.198 [0.156 to 0.252] | 0.286 [0.232 to 0.353]

2. Secondary Outcome: Number of New or Newly Enlarging T2 Hyperintense Lesions
Description: The number of new or newly enlarging T2 hyperintense lesions at 2 years that developed in each subject compared to baseline assessed on brain magnetic resonance imaging (MRI) scans. The estimates of mean T2 hyperintense lesion count were calculated from a negative binomial regression model adjusted for region and baseline T2 hyperintense lesion volume.
Time Frame: 2 years
Population: Of the 681 subjects in the MRI cohort, 572 (139 placebo, 140 BG00012 BID, 140 BG00012 TID, 153 GA) had post-baseline T2 hyperintense data & were included in the analysis. Missing data before the use of alternative MS medications & visits after subjects switched to alternative MS medications were imputed with the use of a constant rate assumption.
Measure: Mean (95% Confidence Interval); unit: Number of lesions
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD)
Number analyzed (Participants) | 139 | 140 | 140 | 153
Number of lesions | 17.4 [13.5 to 22.4] | 5.1 [3.9 to 6.6] | 4.7 [3.6 to 6.2] | 8.0 [6.3 to 10.2]

3. Secondary Outcome: Number of New T1 Hypointense Lesions
Description: The number of new T1 hypointense lesions at 2 years that developed in each subject compared to baseline assessed on brain magnetic resonance imaging (MRI) scans. The estimates of mean T1 hypointense lesion count were calculated from a negative binomial regression model adjusted for region and baseline T1 hypointense lesion volume.
Time Frame: 2 years
Population: Of the 681 subjects in the MRI cohort, 573 (139 placebo,140 BG00012 BID,140 BG00012 TID,154 GA) had post-baseline new T1 hypointense data & were included in the analysis. Missing data before the use of alternative MS medications & visits after subjects switched to alternative MS medications were imputed with the use of a constant rate assumption
Measure: Mean (95% Confidence Interval); unit: Number of lesions
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD)
Number analyzed (Participants) | 139 | 140 | 140 | 153
Number of lesions | 7.0 [5.3 to 9.2] | 3.0 [2.3 to 4.0] | 2.4 [1.8 to 3.2] | 4.1 [3.2 to 5.3]

4. Secondary Outcome: Proportion of Subjects Relapsed
Description: A protocol-defined relapse was defined as new or recurrent neurologic symptoms not associated with fever or infection that lasted at least 24 hours, and were separated by at least 30 days from onset of a preceding relapse. All protocol-defined relapses were evaluated by an independent neurologic evaluation committee. The proportion of subjects with a relapse was estimated using the Kaplan-Meier method, which was based on the time-to-first-relapse survival distribution.
Time Frame: 2 years
Population: The analysis was based on the ITT population, defined as all subjects who were randomized and received at least 1 dose of study treatment. Among subjects who switched to an alternative therapy for MS, all the data before the switch were used for the analysis. In all other subjects, all relapses were included in the analysis.
Measure: Number; unit: Proportion of subjects,confirmed relapse
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD)
Number analyzed (Participants) | 363 | 359 | 345 | 350
Proportion of subjects,confirmed relapse | 0.410 | 0.291 | 0.241 | 0.321

5. Secondary Outcome: Proportion of Subjects Experiencing Progression of Disability Assessed Using the Expanded Disability Status Scale (EDSS)
Description: EDSS is based on a standardized neurological exam and focuses on symptoms that commonly occur in MS. Scores range from 0.0 (normal) to 10.0 (death due to MS). Disability progression was defined as ≥ 1.0 point increase in subjects with a baseline EDSS of ≥1.0, or ≥1.5 point increase in subjects with a baseline EDSS=0, and required that the increase from baseline was confirmed ≥ 12weeks later. The proportion of subjects with confirmed (12-week) disability progression was estimated using the Kaplan-Meier method, which was based on the time-to-first-progression survival distribution
Time Frame: 2 years
Population: The analysis population consisted of the intent-to-treat (ITT) population (all subjects who were randomized and received at least 1 dose of study treatment) who had a baseline EDSS assessment. Analyses were based on all observed data. Onset of disability progression must begin before a subject switched to alternative MS medication.
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD)
Number analyzed (Participants) | 363 | 359 | 345 | 350
Proportion of Participants | 0.169 | 0.128 | 0.130 | 0.156

ADVERSE EVENTS:
Time Frame: 2 years
Description: The safety population consisted of all subjects who received at least 1 dose of study treatment. Safety data were analyzed by actual treatment received. One patient randomly assigned to the BG00012 TID group & included in the group of the ITT population took GA throughout the study and was therefore counted in the GA group of the safety population.
Groups:
- Total BG00012: Combined BG00012 240 mg twice daily (BID) dose group and BG00012 240 mg 3 times daily (TID) dose group
Arm/Group | Placebo | BG00012 240 mg Twice Daily (BID) | BG00012 240 mg 3 Times Daily (TID) | Total BG00012 | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD)
Serious Adverse Events (participants affected / at risk) | 79/363 | 61/359 | 54/344 | 115/703 | 60/351
Other Adverse Events (participants affected / at risk) | 332/363 | 336/359 | 316/344 | 652/703 | 303/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=363) | BG00012 240 mg Twice Daily (BID) (N=359) | BG00012 240 mg 3 Times Daily (TID) (N=344) | Total BG00012 (N=703) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD) (N=351)
GASTROENTERITIS (Infections and infestations) | 0 | 2 | 2 | 4 | 0
CELLULITIS (Infections and infestations) | 0 | 2 | 1 | 3 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 2 | 0
DOUGLAS' ABSCESS (Infections and infestations) | 0 | 0 | 1 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 1 | 1 | 0
H1N1 INFLUENZA (Infections and infestations) | 0 | 1 | 0 | 1 | 0
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 0 | 0 | 1 | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 0 | 1 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 1 | 1
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
BORRELIA INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 2
PYOTHORAX (Infections and infestations) | 0 | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
TRACHEITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
FIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
THYROID CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 0 | 0 | 2
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
BIPOLAR I DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 51 | 39 | 30 | 69 | 36
BENIGN INTRACRANIAL HYPERTENSION (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
DYSARTHRIA (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
GRAND MAL CONVULSION (Nervous system disorders) | 1 | 0 | 1 | 1 | 1
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
MIGRAINE (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
OCCIPITAL NEURALGIA (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
PARTIAL SEIZURES (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
APHASIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
CEREBROVASCULAR DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
CONVULSION (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
EPILEPSY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
EYE PAIN (Eye disorders) | 1 | 0 | 0 | 0 | 0
HOLMES-ADIE PUPIL (Eye disorders) | 1 | 0 | 0 | 0 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 1 | 0 | 0 | 0 | 0
VESTIBULAR ATAXIA (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
MYOCARDITIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0
VOMITING (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
DUODENITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
BLADDER DYSFUNCTION (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
BLADDER PERFORATION (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
BLADDER DIVERTICULUM (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
NEPHROPTOSIS (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 0
GESTATIONAL OEDEMA (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 1
BARTHOLIN'S CYST (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1
ASTHENIA (General disorders) | 1 | 0 | 1 | 1 | 0
HERNIA OBSTRUCTIVE (General disorders) | 0 | 0 | 1 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 1 | 1
PYREXIA (General disorders) | 0 | 0 | 1 | 1 | 0
BETA 2 MICROGLOBULIN URINE INCREASED (Investigations) | 0 | 0 | 1 | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 1
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
EYE INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
WHIPLASH INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
BREAST LUMP REMOVAL (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
INTERVERTEBRAL DISC OPERATION (Surgical and medical procedures) | 0 | 0 | 1 | 1 | 0
MEDICAL DIET (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
CERVICAL CONISATION (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
STERILISATION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
TURBINECTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
SOCIAL PROBLEM (Social circumstances) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=363) | BG00012 240 mg Twice Daily (BID) (N=359) | BG00012 240 mg 3 Times Daily (TID) (N=344) | Total BG00012 (N=703) | Glatiramer Acetate (GA) 20 mg Injection Once Daily (QD) (N=351)
NASOPHARYNGITIS (Infections and infestations) | 58 | 62 | 63 | 125 | 51
URINARY TRACT INFECTION (Infections and infestations) | 42 | 51 | 40 | 91 | 46
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 34 | 36 | 47 | 83 | 27
INFLUENZA (Infections and infestations) | 22 | 20 | 25 | 45 | 15
BRONCHITIS (Infections and infestations) | 14 | 14 | 22 | 36 | 16
SINUSITIS (Infections and infestations) | 11 | 18 | 18 | 36 | 11
DEPRESSION (Psychiatric disorders) | 35 | 24 | 15 | 39 | 28
INSOMNIA (Psychiatric disorders) | 18 | 15 | 10 | 25 | 13
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 147 | 104 | 81 | 185 | 115
HEADACHE (Nervous system disorders) | 49 | 52 | 46 | 98 | 46
PARAESTHESIA (Nervous system disorders) | 31 | 21 | 21 | 42 | 15
HYPOAESTHESIA (Nervous system disorders) | 21 | 11 | 19 | 30 | 16
VERTIGO (Ear and labyrinth disorders) | 22 | 9 | 13 | 22 | 15
FLUSHING (Vascular disorders) | 13 | 110 | 83 | 193 | 6
HOT FLUSH (Vascular disorders) | 8 | 18 | 19 | 37 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 17 | 16 | 18 | 34 | 9
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 | 12 | 21 | 33 | 15
DIARRHEA (Gastrointestinal disorders) | 28 | 45 | 50 | 95 | 14
NAUSEA (Gastrointestinal disorders) | 29 | 40 | 51 | 91 | 15
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 17 | 36 | 33 | 69 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 | 25 | 26 | 51 | 4
VOMITING (Gastrointestinal disorders) | 12 | 25 | 23 | 48 | 8
DYSPEPSIA (Gastrointestinal disorders) | 8 | 12 | 16 | 28 | 6
RASH (Skin and subcutaneous tissue disorders) | 13 | 24 | 28 | 52 | 8
PRURITIS (Skin and subcutaneous tissue disorders) | 11 | 20 | 24 | 44 | 7
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 | 16 | 21 | 37 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 33 | 34 | 36 | 70 | 32
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 26 | 20 | 27 | 47 | 17
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 29 | 21 | 26 | 47 | 21
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 14 | 13 | 21 | 34 | 8
PROTEINURIA (Renal and urinary disorders) | 25 | 29 | 35 | 64 | 30
MICROALBUMINURIA (Renal and urinary disorders) | 13 | 14 | 19 | 33 | 15
FATIGUE (General disorders) | 33 | 37 | 33 | 70 | 30
PYREXIA (General disorders) | 19 | 11 | 24 | 35 | 17
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 0 | 31
INJECTION SITE PAIN (General disorders) | 0 | 0 | 0 | 0 | 29
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 25 | 16 | 22 | 38 | 20
ALBUMIN URINE PRESENT (Investigations) | 15 | 22 | 14 | 36 | 18
PROTEIN URINE PRESENT (Investigations) | 10 | 18 | 7 | 25 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The provisions of our agreement are subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication